CLINICAL TRIAL: NCT03066557
Title: Study of the Combination of Transcatheter Arterial Chemoembolization (TACE) With Apatinib in Patients With Hepatocellular Carcinoma Trial
Brief Title: Study of the Combination of TACE With Apatinib in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shixi Chen, director of department, Jiangsu Cancer Institute & Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANIMATE-JS-201
Record Dates: First submitted 2017-02-20; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Apatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): TACE and Apatinib
  Interventions: Procedure: TACE and Apatinib
- control group (Experimental): TACE alone
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE and Apatinib — TACE and Apatinib 250mg po qd
  Other Names: Aitan
  Arms: study group
Procedure: TACE — TACE
  Arms: control group

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary malignant tumor of the liver. It is lack of effective drugs for systemic treatment of HCC. Currently, Sorafenib is the only choice approved by FDA for advanced HCC, although it prolongs the survival for less than 3 months. The treatment of advanced HCC still has a long way to go.

At present, the relevant phase II and phase III clinical studies of apatinib on advanced HCC are ongoing. Based on our important discovery of previous clinical studies, we intend to enlarge the sample size and make further observation for the efficacy and safety of apatinib in patients with advanced HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the lethal human cancers worldwide and its incidence matches mortality, reflecting the poor prognosis of this disease. The surgical resection rate of HCC is low, and the prognosis is poor. Although transarterial chemoembolization (TACE) is the main treatment for HCC patients who are not candidates for surgical resection, it is not considered a curative procedure. For HCC, poor TACE efficacy or TACE failure may be related to tumor angiogenesis of the residual disease. Among the many regulatory factors in tumor angiogenesis, hypoxia-inducible factor-1α (HIF-1α) and vascular endothelial growth factor (VEGF) play vital roles in this process.

Sorafenib is the first systemic treatment drug, which has been approved by the FDA for advanced HCC. In order to find an new VEGFR-inhibitor with better effect and lower toxicity, Jiangsu Hengrui Medicine Co., Ltd. developed Apatinib, a high-performance VEGFR-2 tyrosine kinase inhibitor. Apatinib plays anti angiogenic effect in the treatment of malignant tumor mainly through inhibition of VEGFR-2, in vivo and in vitro experiments showed good tumor growth inhibitory activity on Hepatocellular carcinoma, this study aims to further verify the efficacy and safety of Apatinib for hepatocellular carcinoma patients who are not candidates for curative surgery, the primary endpoint is Progression Free Survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 75 years old;
2. Must be strictly in accordance with the "guidelines for primary liver cancer diagnosis and treatment" (2011 edition). According to clinical diagnosis standard or confirmed by histopathology or cytology, the patients with advanced primary liver cancer who can't be?removed surgically, and can't accept palliative surgery or radiation therapy, and have at least one measurable lesions;The biggest tumor 10 cm or less;
3. Refuse the treatment of sorafenib;
4. The Child - Pugh( liver function grade): grade A or better grade of B (≤7 points);
5. BCLC stage for B or C;
6. Within 1 week before into the study,ECOG PS0-1;
7. The expected lifetime of patients should be equal to or more than 12 weeks;
8. The main viscera function of patients must be normal, and should meet the following requirements:

   * Blood routine examination must meet: HB≥90 g/L, ANC≥1.5×10^9/L, PLT≥60×10^9/L;
   * Biochemical examination should meet the following criteria: ALB ≥29 g/L, ALT and AST<5xULN, TBIL ≤1.5xULN, creatinine≤1.5xULN (Only one of albumin and bilirubin can be 2 points in the rating of Child-Pugh);
9. The patients are willing to join in this study, and have signed the informed consent. The patients have good adherence, and are willing to cooperate with the follow-up.

Exclusion Criteria:

1. Patients have received radiotherapy or chemotherapy within four weeks before the study;
2. In the past (within 5 years) or at the same time,patients were diagnosed with other malignant tumor which have not been cured. As for skin basal cell carcinoma and cervical carcinoma in situ,they can be excepted;
3. Patients who are diagnosed with hypertension which cant be reduced to normal range via antihypertensive drug treatment(systolic blood pressure> 140 mmHg / diastolic blood pressure> 90 mmHg);
4. Patients who are diagnosed with II or higher level of myocardial ischemia, myocardial infarction, uncontrolled arrhythmia(including QTc interval prolongation men> 450 ms, female> 470 ms);
5. There are many factors which can influence the oral drug absorption (such as unable to swallow, chronic diarrhea and intestinal obstruction, which can significantly affect the drug taking and absorption);
6. Within 6 months in the past,the patients have a history of gastrointestinal bleeding or a gastrointestinal bleeding tendency, for example,there is a risk of bleeding of esophageal varicose veins, local active ulcerative lesions, defecate occult blood ≥ (+ +)(+) shall not be admitted into the study;
7. within 28 days before being admitted into the study, there is abdominal fistula, gastrointestinal perforation or abdominal abscess;
8. Blood coagulation function is abnormal (INR>1.5 or PT> ULN+4s), and the patients are able to be faced with a bleeding tendency or being treated with thrombolysis and anticoagulation;
9. Has been diagnosed with ?the central nervous system metastases or the brain metastases has been known;
10. There are past medical history or history of present illness of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug related pneumonia,pulmonary function test suggests there is objective evidence of severely damaged lung function;
11. Urine routine inspection suggests that the urine protein ≥++;24 hours urine protein examination>1.0 g;
12. Within 7 days before being admitted into the study,patients have received a potent CYP3A4 inhibitor treatment, or within 12 days before being admitted into the study,patients have received potent CYP3A4 inducers treatment;
13. Pregnant or lactating women;Patients with fertility are unwilling or unable to take effective contraceptive measures;
14. With a mental illness, or has a history of psychiatric drugs abuse;
15. Patients with HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-15 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years
  progression free survival

SECONDARY OUTCOMES:
TTP | 2 years
  Time To Progress
OS | 2 years
  Overall Survival
DCR | 2 years
  Disease Control Rate
ORR | 2 years
  Objective Response Rate
QoL | 2 years
  Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Feng Jifeng, Doctor, Study Chair — Jiangsu Cancer Institute & Hospital

IPD SHARING:
Plan to Share IPD: Yes
Within six months after the trial complete